CLINICAL TRIAL: NCT06755723
Title: The Underlying Cause of Mortality and Morbidity in Patients Undergoing Rib Fracture Surgery: Pulmonary Contusion or Associated Extrathoracic Trauma?
Brief Title: Mortality Causes in Rib Surgery Patients
Status: Completed | Type: Observational
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Medical Doctor (MD), Thoracic Surgeon, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/713
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Flail Chest; Rib Fractures; Thoracic Injuries; Pulmonary Contusion; Blunt Trauma
Keywords: Flail chest; Rib fractures; Pulmonary contusion; Multiple trauma
MeSH Terms: conditions — Flail Chest; Rib Fractures; Thoracic Injuries; Wounds, Nonpenetrating; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Rib fractures manangement — This is an observational study, so participants are not assigned interventions. However, the study investigates the outcomes of patients undergoing rib stabilization surgery as part of their routine clinical care. The exposure of interest includes surgical rib stabilization and its timing, combined with any related clinical and care procedures. The outcomes and clinical data collected reflect routine care practices.

SUMMARY:
This study retrospectively investigates the causes of mortality and morbidity in patients undergoing rib fracture surgery due to blunt trauma. The primary objective is to determine whether pulmonary contusion or associated extrathoracic trauma plays a more significant role in adverse outcomes. Data collected includes patient demographics, trauma mechanisms, associated injuries, surgical timing, and clinical outcomes. The study aims to provide insights into improving management strategies for trauma patients and reducing complication rates through early identification and tailored interventions.

DETAILED DESCRIPTION:
This retrospective study investigates the underlying causes of morbidity and mortality in patients who underwent rib stabilization surgery due to blunt trauma-induced rib fractures. The primary objective is to determine whether pulmonary contusion or associated extrathoracic trauma plays a more significant role in adverse outcomes such as pneumonia, prolonged air leaks, tracheostomy, wound infections, and mortality.

The study includes patients diagnosed with flail chest who underwent rib stabilization surgery between January 1, 2014, and January 1, 2024, at a single tertiary care center. Collected data encompasses patient demographics, trauma mechanisms, associated injuries (thoracic and extrathoracic), surgery timing (early vs. late stabilization), ventilator settings, extubation duration, intensive care unit (ICU) and hospital length of stay, laboratory parameters, and clinical outcomes.

Key outcomes include the incidence of morbidity (e.g., pneumonia, prolonged air leak, wound infections) and mortality. Statistical analyses will evaluate the relationship between these outcomes and factors such as the severity and timing of injuries, surgery timing, trauma mechanisms, and associated injuries.

The study aims to provide valuable insights into optimizing the management of flail chest patients, emphasizing the importance of early rib stabilization and a multidisciplinary approach. These findings are expected to contribute to the development of standardized protocols for patient selection and intervention timing, potentially improving patient outcomes in multitrauma settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years diagnosed with flail chest following blunt trauma who underwent rib stabilization surgery
* Those with complete clinical and laboratory data
* Those with at least 30 days of follow-up after surgery.

Exclusion Criteria:

* Patients under 18 years of age
* Flail chest patients who did not require rib stabilization surgery
* Patients with incomplete clinical or laboratory data
* Those with penetrating thoracic trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with blunt trauma-induced rib fractures leading to flail chest, treated with rib stabilization surgery in a hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality Rate in Patients Undergoing Rib Stabilization Surgery | Within 30 days post-surgery
  The primary outcome measure is the overall mortality rate among patients with flail chest due to blunt trauma, treated with rib stabilization surgery. The analysis will focus on the association between mortality and factors such as trauma severity and associated injuries.